CLINICAL TRIAL: NCT03770039
Title: A PHASE 1, OPEN-LABEL, NON-RANDOMIZED, 2-PERIOD, FIXED SEQUENCE STUDY TO INVESTIGATE THE ABSORPTION, DISTRIBUTION, METABOLISM AND EXCRETION OF [14C-PF-06700841] AND TO ASSESS THE ABSOLUTE BIOAVAILABILITY AND FRACTION ABSORBED OF PF-06700841 IN HEALTHY MALE SUBJECTS USING A 14C-MICROTRACER APPROACH
Brief Title: Single Dose Study With Unlabeled Dose and 14C-labeled Microdose of PF-06700841 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7931014; 2018-002403-34 (EudraCT Number)
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Healthy Male Subjects
Keywords: PF-06700841; mass balance; metabolites; absolute bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 2-period, fixed sequence (Experimental): fixed sequence with 2 treatment period
  Interventions: Drug: Oral PF-06700841 containing 14C microtracer; Drug: Oral unlabeled PF-06700841; Drug: IV 14C-labeled PF-06700841

INTERVENTIONS:
Drug: Oral PF-06700841 containing 14C microtracer — Oral dose of 60 mg unlabeled PF-06700841 co-formulated with 30 ug 14C-labeled (300 nCi) PF-06700841 in 1st period
Drug: Oral unlabeled PF-06700841 — 60 mg unlabeled PF-06700841 oral dose in 2nd period
Drug: IV 14C-labeled PF-06700841 — 30 ug 14C-labeled (300 nCi) PF-06700841 intravenous infusion over 5 min in 2nd period

SUMMARY:
An open-label, fixed sequence, 2-period including a single oral dose 60 mg PF-06700841 with 14C-labeled microtracer in 1st period, and a single oral dose of 60 mg unlabeled PF-06700841 followed by intravenous administration of 14C-labeled microdose of PF-06700841 1 hour after oral dose in period 2 to characterize the absorption, disposition, metabolism and excretion of PF-06700841 and evaluate the absolute bioavailability and fraction absorbed in the GI tract

ELIGIBILITY:
Exclusion Criteria:

* Any clinically significant malabsorption condition (eg, gastrectomy, bowel resection).
* Total 14C radioactivity measured in plasma exceeding 11 mBq/mL
* History of tuberculosis or active or latent or inadequately treated infection, positive QuantiFERON®-TB Gold test
* Use of tobacoo/nicotine containing products 3-m prior to dosing or positive urine cotinine test
* Use of herbal supplements within 28 days prior to the first dose of study medication
* Use of prescription or nonprescription drugs (including vitamins and dietary supplements) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. As an exception, acetaminophen may be used at doses of 1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by Pfizer
* Inability to have at least one bowel movement every 2 days on average eGFR of <90 mL/mim/1.73 m2 based on MDRD equation
* Have been vaccinated with live or attenuated live vaccine within the 6 weeks prior to the first dose of investigational product, or expects to be vaccinated with these vaccines during study treatment, or within the 6 weeks following the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
mass balance_urine | hour 0 up to 312 hours post dose
  cumulative recovery of radioactivity over time in urine, as percentage of total radioactive dose administered
mass balance_feces | hour 0 up to 312 hours post dose
  cumulative recovery of radioactivity over time in feces, as percentage of total radioactive dose administered

SECONDARY OUTCOMES:
metabolite identification_plasma | hour 0 up to 312 hours post dose
  metabolic identification and profiling in plasma following a single oral dose of 14C-labeled PF-06700841
plasma Cmax for total 14C radioactivity | hour 0 up to 312 hours post dose
  maximum concentration of total 14C radioactivity in plasma following a single oral dose of 14C-labeled PF-06700841
plasma Tmax for total 14C radioactivity | hour 0 up to 312 hours post dose
  time with highest concentration of radioactivity in plasma following a single oral dose of 14C-labeled PF-06700841
plasma AUClast for total 14C radioactivity | hour 0 up to 312 hours post dose
  area under curve of total 14C radioactivity in plasma from time 0 to tlast following a single oral dose of 14C-labeled PF-06700841
plasma AUCinf for total 14C radioactivity | hour 0 up to 312 hours post dose
  area under curve of total 14C radioactivity in plasma from time 0 to infinite following a single oral dose of 14C-labeled PF-06700841
Oral clearance for total 14C radioactivity | hour 0 up to 312 hours post dose
  oral clearance (CL/F) of total activity following a single oral dose of 14C-labeled PF-06700841
plasma half-life for total 14C radioactivity | hour 0 up to 312 hours post dose
  half-life (t1/2) of total radioactivity in plasma following a single oral dose of 14C-labeled PF-06700841
volume of distribution for total 14C radioactivity | hour 0 up to 312 hours post dose
  apparent volume of distribution (Vz/F) of total radioactivity following a single oral dose of 14C-labeled PF-06700841
plasma Cmax for PF-06700841 | hour 0 up to 96 hours post dose
  maximum concentration of PF-06700841 in plasma following a single oral dose of 14C-labeled or unlabeled PF-06700841
plasma Tmax for PF-06700841 | hour 0 up to 96 hours post dose
  time with highest concentration of PF-06700841 in plasma following a single oral dose of 14C-labeled or unlabeled PF-06700841
plasma AUClast for PF-06700841 | hour 0 up to 96 hours post dose
  area under curve of PF-06700841 in plasma from time 0 to tlast following a single oral dose of 14C-labeled or unlabeled PF-06700841
plasma AUCinf for PF-06700841 | hour 0 up to 96 hours post dose
  area under curve of PF-06700841 in plasma from time 0 to infinite following a single oral dose of 14C-labeled or unlabeled PF-06700841
Oral clearance for PF-06700841 | hour 0 up to 96 hours post dose
  oral clearance (CL/F) of PF-06700841 following a single oral dose of 14C-labeled or unlabeled PF-06700841
plasma half-life for PF-06700841 | hour 0 up to 96 hours post dose
  half-life (t1/2) of PF-06700841 in plasma following a single oral dose of 14C-labeled or unlabeled PF-06700841
volume of distribution for PF-06700841 | hour 0 up to 96 hours post dose
  apparent volume of distribution (Vz/F) of PF-06700841 following a single oral dose of 14C-labeled or unlabeled PF-06700841
plasma Cmax for 14C-labeled PF-06700841 | hour 0 up to 96 hours post dose
  maximum concentration of 14C-labeled PF-06700841 in plasma following a single iv dose of 14C-labeled PF-06700841
plasma Tmax for 14C-labeled PF-06700841 | hour 0 up to 96 hours post dose
  time with highest concentration of 14C-labeled PF-06700841 in plasma following a single iv dose of 14C-labeled PF-06700841
plasma AUClast for 14C-labeled PF-06700841 | hour 0 up to 96 hours post dose
  area under curve of 14C-labeled PF-06700841 in plasma from time 0 to tlast following a single iv dose of 14C-labeled PF-06700841
plasma AUCinf for 14C-labeled PF-06700841 | hour 0 up to 96 hours post dose
  area under curve of 14C-PF-06700841 in plasma from time 0 to infinite following a single iv dose of 14C-labeled PF-06700841
clearance for 14C-labeled PF-06700841 | hour 0 up to 96 hours post dose
  clearance (CL) of 14C-labeled PF-06700841 following a single iv dose of 14C-labeled PF-06700841
plasma half-life for 14C-labeled PF-06700841 | hour 0 up to 96 hours post dose
  half-life (t1/2) of 14C-labeled PF-06700841 in plasma following a single iv dose of 14C-labeled PF-06700841
volume of distribution for 14C-labeled PF-06700841 | hour 0 up to 96 hours post dose
  volume of distribution (Vz/F) of 14C-labeled PF-06700841 following a single iv dose of 14C-labeled PF-06700841
unchanged PF-06700841 recovered in urine | hour 0 up to 96 hours post dose
  percentage of unchanged PF-06700841 recovered in urine (Ae%) following a single oral dose of PF-06700841
renal clearance of PF-06700841 | hour 0 up to 96 hours post dose
  renal clearance (CLr) following a single oral dose of PF-06700841 (Ae%/AUCinf for PF-06700841)
Bioavailability of oral PF-06700841 | hour 0 up to 96 hours post dose
  Absolute bioavailability (F) following a single oral dose relative to a single iv dose of PF-06700841
Fraction absorbed of oral PF-06700841 | hour 0 up to 144 hours post dose
  Fraction absorbed in gut (Fa) following oral dose of PF-06700841
metabolite identification_urine | hour 0 up to 312 hours post dose
  metabolic identification and profiling in urine following a single oral dose of 14C-labeled PF-06700841
metabolite identification_feces | hour 0 up to 312 hours post dose
  metabolic identification and profiling in feces following a single oral dose of 14C-labeled PF-06700841

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Netherlands (2):
  - PRA Health Sciences, Groningen
  - PRA Health Sciences Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Qiu R, Sharma R, Wei H, Kirkovsky L, Zhou Y, Martin DDA, Banfield C, Dowty ME. A phase 1 study to investigate the absorption, distribution, metabolism and excretion of brepocitinib in healthy males using a 14 C-microdose approach. Br J Clin Pharmacol. 2023 Oct;89(10):3056-3066. doi: 10.1111/bcp.15786. Epub 2023 Jun 20. PMID 37183779
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7931014&StudyName=A+Phase+1%2C+Open-label%2C+Non-randomized%2C+2-period%2C+Fixed+Sequence+Study+To+Investigate+The+Absorption%2C+Distribution%2C+Metabolism+And+Excretion+Of+%5B14c-pf-06700841%5D+And+To+Assess+The+Absolute+Bioavailability+And+Fraction+Absorbed+Of+Pf-06700841+In+Healthy+Male+Subjects+Using+A+14c-microtracer+Approach